CLINICAL TRIAL: NCT06362993
Title: Testing Approaches to Promote Breast Cancer Screening in Rural Ghana
Brief Title: Breast Cancer Screening in Ghana
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: University of Ghana (Other)
Responsible Party: Principal Investigator, Yubraj Acharya, Ph.D., Associate Professor, Penn State University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: STUDY00021561
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Women in this arm receive education on breast cancer and are offered clinical breast exam free of charge at their local clinic for 6 months following the education session.
- Bundling (Experimental): Women in this arm receive education on breast cancer, diabetes, and hypertension, and are offered clinical breast exam and screening for diabetes and hypertension free of charge at their local clinic for 6 months following the education session.
  Interventions: Other: Bundling
- Male Engagement in Gender and Health (MEGH) (Experimental): Women in this arm receive education on breast cancer and are offered clinical breast exam free of charge at their local clinic for 6 months following the education session. In addition, women are requested to invite their male partners to attend the breast cancer education session and 7 weekly discussion group sessions (5 men-only and 2 with women). The discussion sessions aim to enable men to change gender attitudes and behaviors that deter women's healthcare utilization.
  Interventions: Other: MEGH

INTERVENTIONS:
Other: Bundling — Education on and screening for diabetes and hypertension offered together with education and screening for breast cancer.
  Arms: Bundling
Other: MEGH — Education on breast cancer and discussion sessions to male partners to change men's gender attitudes and behaviors.
  Arms: Male Engagement in Gender and Health (MEGH)

SUMMARY:
This study is designed to test the feasibility of two intervention on promoting early screening for breast cancer in rural Ghana. In one intervention, screening for breast cancer, diabetes and hypertension will be offered together. In another intervention, a series of sessions with men will be conducted with a goal to change gender attitudes and increase support to women. The investigators' long-term goal is to test these interventions in a large-scale randomized controlled trial. The specific aims of this feasibility study are to: 1) refine the study materials, including the curriculum for the sessions with men, by consulting with an expert advisory committee and a local committee, and 2) determine the feasibility of the two interventions in four clinic zones in Yilo-Krobo district in eastern Ghana (1 clinic in control, 1 clinic in the first intervention, and 2 in the second intervention). This trial registration is for the second specific aim.

ELIGIBILITY:
Inclusion Criteria:

* ≥20 years. The age cutoff reflects early onset of BC in Ghana and the government's guidelines on screening.

Exclusion Criteria:

* ever clinically diagnosed with a case of breast cancer, as the study's aim is to reach women who would normally not visit or have experience with the health system with regard to breast cancer.

NOTE: For men in the MEGH arm, Inclusion and Exclusion Criteria are:

Inclusion Criteria: aged ≥20 years who are identified as male partners or relatives by the women enrolled in the MEGH group.

Exclusion Criteria: none.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2024-08-18 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Clinical breast exam (CBE) utilization at the local clinic | 6 months. Outcome is measured at endline survey at the end of the 6-month period.
  The outcome will be measured by asking participants, at endline, if they sought clinical breast exam at their local clinic during the 6-month study period. This information will be verified at the clinic level using Participation Cards, which will be provided to participants at the beginning of the 6-month period. Participants will be asked to bring the Card to the clinic when they come for screening.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Luke, Ph.D., Study Chair — The Pennsylvania State University; Adriana Biney, Ph.D., Study Chair — University of Ghana, Regional Institute for Population Studies
Locations (1):
- University of Ghana, Accra, Ghana